CLINICAL TRIAL: NCT02625623
Title: A Phase III Open-label, Multicenter Trial of Avelumab (MSB0010718C) as a Third-line Treatment of Unresectable, Recurrent, or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Avelumab in Third-Line Gastric Cancer (JAVELIN Gastric 300)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 100070-008; 2015-003301-42 (EudraCT Number)
Record Dates: First submitted 2015-12-04; First posted 2015-12-09 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-10

CONDITIONS: Unresectable, Recurrent, Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma; Gastric Cancer Third Line
Keywords: Avelumab; Gastric cancer; Gastroesophageal junction adenocarcinoma
MeSH Terms: conditions — Recurrence; Stomach Neoplasms | interventions — avelumab; Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Physician choice chemotherapy+Best Supportive Care (BSC) (Experimental): Participants received BSC plus physician's choice chemotherapy. Chemotherapy comprises of one of the following: paclitaxel at a dose of 80 milligram per meter square (mg/m^2) on Days 1, 8, and 15 of a 4-week treatment cycle until confirmed progressive disease or unacceptable toxicity OR irinotecan at a dose of 150 mg/m^2 on Days 1 and 15 of a 4-week treatment cycle until confirmed progressive disease or unacceptable toxicity. Participants who are not deemed eligible to receive paclitaxel or irinotecan at the dose and schedule specified above receive BSC alone once every 3 weeks. BSC is defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and is based on investigator's discretion.
  Interventions: Drug: Irinotecan; Drug: Paclitaxel; Other: Best Supportive Care (BSC)
- Avelumab+BSC (Active Comparator): Participants received avelumab as a 1-hour intravenous (IV) infusion at 10 milligram per kilogram (mg/kg) once every 2-week treatment cycle until confirmed progressive disease or unacceptable toxicity along with BSC. BSC is defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and is based on investigator's discretion.
  Interventions: Drug: Avelumab; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Avelumab — Avelumab was administered as a 1-hour intravenous (IV) infusion at 10 milligram per kilogram (mg/kg) once every 2-week treatment cycle until confirmed progressive disease or unacceptable toxicity along with best supportive care (BSC).
  Other Names: MSB0010718C; Anti PD-L1
  Arms: Avelumab+BSC
Drug: Irinotecan — Irinotecan was administered at a dose of 150 mg/m ^2 on Day 1 and 15 of a 4-week treatment cycle until disease progression or unacceptable toxicities along with BSC.
  Arms: Physician choice chemotherapy+Best Supportive Care (BSC)
Drug: Paclitaxel — Paclitaxel was administered at a dose of 80 mg/m^2 on Day 1, 8, and 15 of a 4-week treatment cycle until disease progression or unacceptable toxicities along with BSC.
  Arms: Physician choice chemotherapy+Best Supportive Care (BSC)
Other: Best Supportive Care (BSC) — BSC is defined as treatment administered with the intent to maximize Quality of life without a specific antineoplastic regimen and is based on investigator's discretion. BSC was administered once every 3 weeks.

SUMMARY:
The purpose of this study was to demonstrate superiority of treatment with avelumab plus best supportive care (BSC) versus physician's choice (chosen from a pre-specified list of therapeutic options) plus BSC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged greater than or equal to (>=) 18 years
* Subjects with histologically confirmed recurrent unresectable, recurrent locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction (GEJ)
* Availability of a formalin-fixed, paraffin-embedded (FFPE) block containing tumor tissue
* Subjects must have received 2 prior courses of systemic treatment for unresectable, recurrent, locally advanced or metastatic gastric cancer, and must have progressed after the second line
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1 at trial entry
* Adequate hematological, hepatic and renal functions defined by the protocol
* Negative blood pregnancy test at Screening for women of childbearing potential.
* Highly effective contraception for both male and female subjects if the risk of conception exists

Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Prior therapy with any antibody or drug targeting T-cell coregulatory proteins
* Concurrent anticancer treatment
* Major surgery
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to less than [<] 10 mg prednisone daily).
* All subjects with brain metastases, except those meeting the following criteria: a. Brain metastases have been treated locally, and b. No ongoing neurological symptoms that are related to the brain localization of the disease (sequelae that are a consequence of the treatment of the brain metastases are acceptable)
* Previous malignant disease (other than gastric cancer) within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or carcinoma in situ (bladder,cervical, colorectal, breast)
* Prior organ transplantation, including allogeneic stem-cell transplantation Significant acute or chronic infections
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Persisting toxicity of grade >2 related to prior therapy except neuropathy and alopecia
* Neuropathy Grade greater than or equal (>=) 3.
* Pregnancy or lactation
* Known alcohol or drug abuse
* History of uncontrolled intercurrent illness including hypertension, active infection, diabetes
* Clinically significant (i.e., active) cardiovascular disease
* All other significant diseases might impair the subject's tolerance of trial treatment
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent and that would limit compliance with study requirements
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines
* Legal incapacity or limited legal capacity
* Subjects will be excluded from the treatment with irinotecan or paclitaxel monotherapy if administration of their chemotherapy would be inconsistent with the current local labeling (for example, in regard to contraindications, warnings/precautions, or special provisions) for that chemotherapy. Investigators should check updated labeling via relevant websites before randomization
* Subjects should start treatment administration within 28 days after signing the informed consent form (ICF). Treatment administration will start within 4 days after the randomization call

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (75):
- United States (28):
  - Rocky Mountain Cancer Centers 1800 Williams Street, Suite 100, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP 3676 Parker Blvd #350, Pueblo, Colorado
  - Advanced Medical Specialties 8940 North Kendall Drive, Suite 300E, Miami, Florida
  - Ocala Oncology Center, P.L. 433 S.W. 10th Street, Ocala, Florida
  - Florida Cancer Specialists 560 Jackson Street, Suite 220, St. Petersburg, Florida
  - Ingalls Memorial Hospital One Ingalls Drive, W741, Harvey, Illinois
  - Illinois Cancer Specialists 8915 W. Golf Rd., Niles, Illinois
  - Oncology Specialists, S.C. 1700 Luther Ln, Ste 2200, Park Ridge, IL 60068 7900 Milwaukee Ave, Ste 16, Niles, Illinois
  - Carle Cancer Center 509 W. University Avenue, Urbana, Illinois
  - Cotton-O'Neil Clinical Research Center, Hematology and Oncology and Stormont Vail Cancer Center 1414 SW 8th St, Topeka, Kansas
  - Metairie Oncologist, LLC Office of Jayne Gurtler MD, Laura Brinz MD, Janet Burroff MD 3939 Houma Blvd, Suite 6, Metairie, Louisiana
  - Henry Ford Health System 2799 West Grand Boulevard, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A. 910 East 26th Street, Suites 100 and 200, Minneapolis, Minnesota
  - Southern Nevada Cancer Research Foundation 601 S Rancho Drive, Las Vegas, Nevada
  - New York Oncology Hematology, P.C. 400 Patroon Creek Blvd, Suite 1, Albany, New York
  - Sanford Roger Maris Cancer Center - Fargo 801 Broadway North Route 1058, Fargo, North Dakota
  - Northwest Cancer Specialists, P.C. 265 N Broadway, Portland, Oregon
  - Penn State University Milton S. Hershey Medical Center 500 University Drive, Hershey, Pennsylvania
  - Hematology and Oncology Associates of SC, LLC 900 West Faris Rd, 3rd Floor, Greenville, South Carolina
  - Tennessee Oncology 250 20th Ave North, Nashville, Tennessee
  - Texas Oncology Bedford 1609 Hospital Parkway, Bedford, Texas
  - Texas Oncology, P.A. 3410 Worth Street, Suites 300 & 400, Dallas, Texas
  - Texas Oncology, P.A. - Denton 3720 South I-35 East, Denton, Texas
  - Oncology Consultants, P.A. 2130 W. Holcombe Blvd. 10th Floor, Houston, Texas
  - Texas Oncology, P.A. - McAllen 1901 South 2nd Street, McAllen, Texas
  - Scott and White Memorial Hospital and Clinic 2401 South 31st Street, Temple, Texas
  - Texas Oncology, P.A. - Tyler 910 E. Houston St, Suite 100, Tyler, Texas
  - Texas Oncology - Waco 1700 W. Hwy. 6, Waco, Texas
- Australia (8):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Fiona Stanley Hospital, Subiaco, Western Australia
- Belgium (8):
  - OLV Ziekenhuis, Aalst
  - AZ Sint Lucas, Bruges
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - CHC Clinique StJospeh, Liège
  - CHU Sart Tilman, Liège
  - AZ Turnhout - Campus Sint-Elisabeth, Turnhout
- Nemocnice Rudolfa a Stefanie Benesov, a. s., Benešov, Czechia
- France (3):
  - Service d'Oncologie Médicale, Brest, Finistere
  - Service d'Hépato-Gastro-Entérologie, La Roche S/ Yon Cedex 9, Vendee
  - Centre Oscar Lambret, Lille
- Germany (5):
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Schwerpunktpraxis für Haematologie und Onkologie, Magdeburg, Saxony-Anhalt
  - Charite Universitaetsmedizin, Berlin
  - Schwerpunktpraxis für Haematologie und OnkologieOnkologische Schwerpunktpraxis Eppendorf, Hamburg
  - Leopoldina Krankenhaus, Schweinfurt
- Italy (3):
  - A.O.U. Ospedali Riuniti Ancona- Clinica Oncologica, Torrette Di Ancona, Ancona
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Ospedale San Raffaele, Milan
- Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw, Poland
- South Korea (10):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-Gun, Jeollanam-do
  - Kyungpook National University Medical Center, Daegu
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Seoul National Univ Hospital, Seoul
- Spain (8):
  - Hospital Univ Vall dHebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinico San Carlos Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario la Paz - site 546, Madrid
  - Hosp Univer Madrid Sanchinarro, Madrid

REFERENCES:
- [Result] Bang YJ, Ruiz EY, Van Cutsem E, Lee KW, Wyrwicz L, Schenker M, Alsina M, Ryu MH, Chung HC, Evesque L, Al-Batran SE, Park SH, Lichinitser M, Boku N, Moehler MH, Hong J, Xiong H, Hallwachs R, Conti I, Taieb J. Phase III, randomised trial of avelumab versus physician's choice of chemotherapy as third-line treatment of patients with advanced gastric or gastro-oesophageal junction cancer: primary analysis of JAVELIN Gastric 300. Ann Oncol. 2018 Oct 1;29(10):2052-2060. doi: 10.1093/annonc/mdy264. PMID 30052729
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR%20100070-008
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 459 participants were screened for this study. Of which, 371 participants were randomized into the study.
Groups:
- Physician Choice Chemotherapy + Best Supportive Care (BSC): Participants received BSC plus physician's choice chemotherapy. Chemotherapy comprised of one of the following: intravenous (IV) infusion of paclitaxel at a dose of 80 milligrams per meter square (mg/m^2) on Days 1, 8 and 15 of a 4-week treatment cycle until progressive disease or unacceptable toxicity OR irinotecan at a dose of 150 mg/m^2 on Days 1 and 15 of a 4-week treatment cycle until progressive disease or unacceptable toxicity. Participants who were not deemed eligible to receive paclitaxel or irinotecan at the dose and schedule specified above received BSC alone once every 3 weeks. BSC was defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and was based on investigator's discretion.
- Avelumab + BSC: Participants received avelumab as a 1-hour intravenous (IV) infusion at 10 milligrams per kilogram (mg/kg) once every 2-week treatment cycle until progressive disease or unacceptable toxicity along with BSC. BSC was defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and was based on investigator's discretion.
Period: Overall Study
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Started | 186 | 185
Treated | 177 | 184
Completed | 177 | 184
Not Completed | 9 | 1
Not completed — Participants randomized but not treated | 9 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC | Total
Number analyzed (Participants) | 186 | 185 | 371
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (12.93) | 58.8 (11.66) | 59.5 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 45 | 104
  Male | 127 | 140 | 267
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 15 | 30
  Not Hispanic or Latino | 150 | 153 | 303
  Unknown or Not Reported | 21 | 17 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 117 | 119 | 236
  Black or African American | 1 | 1 | 2
  Asian | 47 | 47 | 94
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Not collected/Missing | 19 | 15 | 34
  Other | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. For participants who were still alive at the time of data analysis or who were lost to follow-up, OS time was censored at the date of last contact. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: From randomization up to 627 days
Population: FAS included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 186 | 185
months | 5.0 [4.5 to 6.3] | 4.6 [3.6 to 5.7]
Statistical Analysis 1: Comparison: Physician Choice Chemotherapy + Best Supportive Care (BSC) vs Avelumab + BSC; Test type: Superiority; p = 0.8078, Log Rank; The treatment arms were compared using a stratified, 1-sided, log rank Test. The stratification factor was region (Asia versus non Asia); Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.88 to 1.41]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS time was defined as the time from date of randomization until date of the first documentation of progressive disease (PD) or death due to any cause (whichever occurs first). PFS was assessed as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: From randomization up to 627 days
Population: FAS included all participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 186 | 185
months | 2.7 [1.81 to 2.83] | 1.4 [1.38 to 1.45]
Statistical Analysis 1: Comparison: Physician Choice Chemotherapy + Best Supportive Care (BSC) vs Avelumab + BSC; Test type: Superiority; p = 1.0000, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [1.36 to 2.21]

3. Secondary Outcome: Best Overall Response (BOR)
Description: BOR was determined by RECIST v1.1 and defined as best-confirmed response of any of following: complete response (CR), partial response (PR), stable disease (SD) and PD recorded from date of randomization until disease progression or recurrence. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in SLD of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD is defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or appearance of 1 or more new lesions. PR or CR confirmed at a subsequent tumor assessment, not sooner than 5 weeks after initial documentation or at an assessment later than the next assessment after the initial documentation of PR or CR. SD confirmed at least 6 weeks after randomization. Confirmed PD equal to progression <=2 weeks after date of randomization (and not qualifying for CR, PR or SD).
Time Frame: From randomization up to 627 days
Population: FAS included all participants who were randomized to study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Avelumab + BSC: Participants received avelumab as a 1-hour intravenous (IV) infusion at 10 milligram per kilogram (mg/kg) once every 2-week treatment cycle until progressive disease or unacceptable toxicity along with BSC. BSC was defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and was based on investigator's discretion.
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 186 | 185
Participants
  Complete Response | 1 | 1
  Partial response | 7 | 3
  Stable disease | 62 | 30
  Non-complete response/ Non-progressive disease | 12 | 7
  Progressive disease | 59 | 94
  Non-evaluable | 45 | 50

4. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR defined as the percentage of all randomized participants with a confirmed best overall response (BOR) of partial response (PR),or complete response (CR) according to RECIST v1.1 and as adjudicated by the Independent Review Committee (IRC). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions.
Time Frame: From randomization up to 627 days
Population: FAS included all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Avelumab + SC: Participants received avelumab as a 1-hour intravenous (IV) infusion at 10 milligram per kilogram (mg/kg) once every 2-week treatment cycle until progressive disease or unacceptable toxicity along with BSC. BSC was defined as treatment administered with the intent to maximize quality of life without a specific antineoplastic regimen and was based on investigator's discretion.
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + SC
Number analyzed (Participants) | 186 | 185
percentage of participants | 4.3 [1.9 to 8.3] | 2.2 [0.6 to 5.4]
Statistical Analysis 1: Comparison: Physician Choice Chemotherapy + Best Supportive Care (BSC) vs Avelumab + SC; Test type: Superiority; p = 0.8764, Cochran-Mantel-Haenszel; The treatment arms were compared by 1-sided CMH test. The stratification factor was region (Asia versus non Asia); Odds Ratio (OR) = 0.709

5. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire Through Composite Index Score at End of Treatment (EOT)
Description: EQ-5D-5L is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive overall composite health state index score, with scores ranging from -0.594 to 1. A higher score indicates better health state.
Time Frame: Baseline, EOT (up to Week 66)
Population: Health-related quality of life (HRQoL) analysis set included a subset of the FAS and included FAS participants who met the following criteria: had 1 Baseline HRQoL assessment, had at least 1 post-Baseline HRQoL questionnaire completed. "Number of Participants Analyzed" signifies the number of participants analyzed in this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 92 | 74
units on a scale | -0.103 (0.2113) | -0.144 (0.2088)

6. Secondary Outcome: Change From Baseline in European Quality of Life 5-dimensions (EQ-5D-5L) Health Outcome Questionnaire Through Visual Analogue Scale (VAS) at End of Treatment (EOT)
Description: EQ-5D-5L is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
Time Frame: Baseline, EOT (up to Week 66)
Population: HRQoL analysis set included a subset of the FAS and included FAS participants who met the following criteria: had 1 Baseline HRQoL assessment, had at least 1 post-Baseline HRQoL questionnaire completed. "Number of Participants Analyzed" signifies the number of participants analyzed in this outcome.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 92 | 74
millimeter (mm) | -12.3 (19.22) | -13.6 (19.76)

7. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status Scale Score at End of Treatment (EOT)
Description: EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnoea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact. The EORTC QLQ-C30 GHS/QoL score ranges from 0 to 100; High score indicates better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Time Frame: Baseline, EOT (up to Week 66)
Population: HRQoL analysis set included a subset of the FAS and included FAS participants who met the following criteria: had 1 Baseline HRQoL assessment and had at least 1 post-Baseline HRQoL questionnaire completed. "Number of Participants Analyzed" signifies the number of participants analyzed in this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 92 | 74
units on a scale | -10.14 (19.914) | -15.77 (19.437)

8. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Stomach Cancer Specific (EORTC QLQ-STO22) Questionnaire Scores at End of Treatment (EOT)
Description: The EORTC QLQ-STO22 supplements the EORTC QLQ-C30 to assess symptoms and treatment-related side effects commonly reported in participants. There are 22 questions which comprise 5 scales (dysphagia, pain, reflux symptom, dietary restrictions, and anxiety) and 4 single items (dry mouth, hair loss, taste, body image). Most questions use 4-point scale (1 'Not at all' to 4 'Very much'; 1 question was a yes or no answer). A linear transformation was used to standardize all scores and single-items to a scale of 0 to 100; higher score=better level of functioning or greater degree of symptoms.
Time Frame: Baseline, EOT (up to Week 66)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
Number analyzed (Participants) | 92 | 74
units on a scale
  Dysphagia | 7.25 (28.551) | 15.32 (29.120)
  Pain | 8.88 (22.402) | 9.23 (21.527)
  Reflux | 4.59 (20.184) | 7.96 (18.347)
  Eating Restrictions | 9.24 (22.661) | 13.29 (21.276)
  Anxiety | 7.49 (21.860) | 6.61 (19.456)
  Dry Mouth | 15.94 (27.725) | 9.01 (28.827)
  Tasting | 9.42 (25.832) | 2.25 (35.897)
  Body Image | 5.07 (28.787) | 4.05 (27.561)
  Hair Loss | 4.71 (33.546) | -13.96 (26.029)

ADVERSE EVENTS:
Time Frame: From randomization up to 627 days
Description: All participants who received at least 1 dose of study drug (that is, treated participants) were included in safety population.
Arm/Group | Physician Choice Chemotherapy + Best Supportive Care (BSC) | Avelumab + BSC
All-Cause Mortality (participants affected / at risk) | 131/177 | 142/184
Serious Adverse Events (participants affected / at risk) | 81/177 | 90/184
Other Adverse Events (participants affected / at risk) | 150/177 | 146/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Physician Choice Chemotherapy + Best Supportive Care (BSC) (N=177) | Avelumab + BSC (N=184)
Disease progression (General disorders) | 30 | 39
General physical health deterioration (General disorders) | 3 | 11
Asthenia (General disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 6
Vomiting (Gastrointestinal disorders) | 1 | 5
Intestinal obstruction (Gastrointestinal disorders) | 1 | 4
Ascites (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 3
Ileus (Gastrointestinal disorders) | 4 | 2
Subileus (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Pneumonia (Infections and infestations) | 2 | 5
Sepsis (Infections and infestations) | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Condition aggravated (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Sudden death (General disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Liver function test increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Autoimmune hypothyroidism (Endocrine disorders) | 0 | 1
Device occlusion (Product Issues) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Shock symptom (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Physician Choice Chemotherapy + Best Supportive Care (BSC) (N=177) | Avelumab + BSC (N=184)
Nausea (Gastrointestinal disorders) | 61 | 34
Vomiting (Gastrointestinal disorders) | 32 | 33
Abdominal pain (Gastrointestinal disorders) | 31 | 25
Diarrhoea (Gastrointestinal disorders) | 54 | 24
Constipation (Gastrointestinal disorders) | 27 | 18
Dysphagia (Gastrointestinal disorders) | 2 | 10
Abdominal pain upper (Gastrointestinal disorders) | 18 | 7
Fatigue (General disorders) | 28 | 28
Asthenia (General disorders) | 35 | 26
Pyrexia (General disorders) | 30 | 21
Chills (General disorders) | 3 | 19
Oedema peripheral (General disorders) | 16 | 5
Aspartate aminotransferase increased (Investigations) | 13 | 16
Weight decreased (Investigations) | 12 | 16
Gamma-glutamyltransferase increased (Investigations) | 13 | 15
Blood alkaline phosphatase increased (Investigations) | 10 | 14
Alanine aminotransferase increased (Investigations) | 13 | 11
Neutrophil count decreased (Investigations) | 16 | 0
White blood cell count decreased (Investigations) | 14 | 0
Decreased appetite (Metabolism and nutrition disorders) | 37 | 29
Dehydration (Metabolism and nutrition disorders) | 3 | 10
Anaemia (Blood and lymphatic system disorders) | 48 | 30
Neutropenia (Blood and lymphatic system disorders) | 25 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT02625623/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT02625623/SAP_003.pdf